CLINICAL TRIAL: NCT07106788
Title: Aveir Leadless Pacemaker Japan Post Marketing Surveillance
Brief Title: Aveir Leadless Pacemaker Japan PMS
Status: Recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CL1027565
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Leadless Pacemaker
Keywords: leadless pacemaker; AVEIR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (4):
- Primary Analysis Cohort: This survey targets the registration of 194 patients indicated for de novo dual-chamber LP's. All de novo patients will be followed until the last de novo dual-chamber patient (Aveir Japan PMS primary analysis cohort) reaches 3 years of follow-up
  Interventions: Device: Aveir DR Leadless Pacemaker Implant
- Single-chamber atrial Aveir patients: Up to 50 patients indicated for a de novo atrial LP may be registered during the primary de novo dual-chamber LP registration period. Data will be analyzed separately, and the patients will be followed until the last de novo dual-chamber patient (primary analysis cohort) reaches 3 years of follow-up
  Interventions: Device: Single-chamber atrial Aveir patients
- Upgrade Patients: Up to 36 upgrade patients (existing ventricular LP to dual-chamber LP system or existing atrial LP to dual-chamber LP system) may be registered during the primary de novo dual-chamber LP registration period. Data will be analyzed separately, and the patients will be followed until the last de novo dual-chamber patient (primary analysis cohort) reaches 3 years of follow-up
  Interventions: Device: Upgrades
- Rollover: All patients from Japan sites with existing active Aveir LPs from the Aveir DR IDE i2i Study (up to 24 patients) are eligible to roll over into the Aveir Japan PMS upon consent for ongoing follow-up. Data from the rollover patients will be summarized separately. Rollover patients will be followed until the last de novo dual-chamber patient (Aveir Japan PMS primary analysis cohort) reaches 3 years of follow-up
  Interventions: Device: Roll-over

INTERVENTIONS:
Device: Aveir DR Leadless Pacemaker Implant — Patients will undergo a dual chamber leadless pacemaker system implant wherein a leadless pacemaker will be implanted in the right ventricle and right atrium
  Groups: Primary Analysis Cohort
Device: Single-chamber atrial Aveir patients — Patients will undergo a single chamber leadless pacemaker system implant wherein a leadless pacemaker will be implanted in the right atrium
  Groups: Single-chamber atrial Aveir patients
Device: Upgrades — Patients with an existing single-chamber leadless pacemaker will undergo a leadless pacemaker system implant wherein an additional leadless pacemaker will be implanted in either the right ventricle or right atrium to form a dual-chamber LP system.
  Groups: Upgrade Patients
Device: Roll-over — Patients with an existing active Aveir DR leadless pacemaker system are eligible to be rolled into the Aveir Japan PMS upon consent for ongoing follow-up.
  Groups: Rollover

SUMMARY:
The primary purpose of the PMS is to collect safety information on the Aveir DR leadless cardiac pacemaker (LP) system in a population indicated for de novo dual-chamber pacing. Additionally, the PMS will collect data on rollover patients from the Aveir DR i2i IDE, Aveir AR LP in patients indicated for single-chamber pacing in the right atrium, and upgradeability in patients implanted with single-chamber Aveir atrial or ventricular LP that require an upgrade to a dual-chamber Aveir LP.

ELIGIBILITY:
Inclusion Criteria:

* Patient is indicated for dual-chamber or single-chamber atrial leadless pacemaker system
* Patient is a roll-over patient with existing Aveir DR leadless pacemaker system from the Aveir DR i2i IDE study
* Patient is an upgrade patient with existing single-chamber Aveir leadless pacemaker that requires an upgrade to a dual-chamber Aveir leadless pacemaker system

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Surveillance will register patients who are indicated for dual-chamber leadless pacemaker, single-chamber atrial leadless pacemaker, roll-over patients with existing Aveir DR leadless pacemaker system from the Aveir DR i2i IDE study, and upgrade patients with existing single-chamber Aveir leadless pacemaker that require an upgrade to a dual-chamber Aveir leadless pacemaker system.
Sampling Method: Non-Probability Sample
Enrollment: 304 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 36-month
  The primary safety endpoint of this PMS evaluates the 3-year Aveir DR LP system complication-free rate in de novo Aveir DR patients (primary analysis group).
  A complication is defined as a device-or-procedure-related serious adverse device effect (SADE), including those that prevent initial implantation (includes both Atrial LP and Ventricular LP related complications and implant procedure-related complications).

OTHER OUTCOMES:
Key Survey Items - Descriptive Endpoints | 36-month
  The key survey item - descriptive endpoints are evaluated as rates for the following adverse events for all patients:
  * Atrial fibrillation
  * Dislodgement of atrial LP
  * Myocardial injury (defined as cardiac perforation, pericardial effusion, or cardiac tamponade)
  * Physical interference with other procedures or devices
  Additionally, the number of events of atrial LP removal and the success rate of removals will be reported.

CONTACTS AND LOCATIONS:
Locations (9):
- Japan (9):
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagwa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Osaka Keisatsu Hospital, Osaka, Osaka
  - National Cerebral & Cardiovascular Center Hospital, Suita, Osaka
  - Juntendo University Shizuoka Hospital, Izunokuni, Shizuok
  - Tokyo Medical University Hospital, Tokyo, Tokyo
  - Tokyo Women's Hospital, Tokyo, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Any de-identified individual participant data collected will be shared with investigators whose proposed use of the data has been approved by Abbott
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be available following publication of primary results for 25 years following study completion date.
Access Criteria: Proposals for requesting individual data may be submitted to the Sponsor at AveirDR_IDE@abbott.com.